CLINICAL TRIAL: NCT03574389
Title: A PHASE 3 OPEN-LABEL TRIAL TO ASSESS THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF 13-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN INFANTS AND YOUNG CHILDREN IN CHINA WHO ARE NAIVE TO PNEUMOCOCCAL VACCINATION
Brief Title: A Study Assessing 13-valent Pneumococcal Conjugate Vaccine in Healthy Chinese Infants and Young Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B1851178
Record Dates: First submitted 2018-05-22; First posted 2018-07-02 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Pneumococcal Infections; Pneumococcal Conjugate Vaccine
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 13-valent Pneumococcal Conjugate Vaccine (13vPnC) (Experimental): 1. Participants in cohort 1 will receive each dose of 13vPnC in months 2, 4 and 6, and then a booster dose during months 12-15.
  2. Participants in cohort 2 will receive first dose dose 13vPnC at the age of months 7(included) to months 12 (less than months 12), and the second dose will be given at least 28 days after first dose, and the third dose will be months 12 to 15 (and at least 56 days after the second dose).
  3. Participants in cohort 3 will receive the first dose of 13vPnC during 1 (included) to 2 years (less than 2 years of age) of age, and the second dose will be given at least 56 days after first dose.
  4. Participants in cohort 4 will receive only one dose at the age of 2 (included) to 6 (less than 6 years of age) years of age.
  Interventions: Biological: 13vPnC
- Haemophilus influenzae type b (Hib) (Active Comparator): 1. No participants in cohort 1 will receive Hib vaccine.
  2. Participants in cohort 2 will receive the first dose of Hib vaccine at the age of months 7 (included) to 12 (less than 12 months), and the second dose will be given at least 28 days after the first dose, the third dose will following local practice or national recommendation at the discretion of the investigator.
  3. Participants in cohorts 3 and 4 will receive the only one dose Hib vaccine at the age of 1 (included) to 6 (less than 6 years) years of age.
  Interventions: Biological: Hib

INTERVENTIONS:
Biological: 13vPnC — suspension in prefilled syringe for intramuscular injection, 0.5 mL, only one dose
  Arms: 13-valent Pneumococcal Conjugate Vaccine (13vPnC)
Biological: Hib — suspension in prefilled syringe for intramuscular injection, 0.5 mL, only one dose
  Arms: Haemophilus influenzae type b (Hib)

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of 13-valent Pneumococcal conjugate vaccine in Chinese infant and young children.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated ICD indicating that the parent(s)/legal guardian has been informed of all pertinent aspects of the study.
* Aged 6 weeks (42 days) to <6 years at the time of consent.
* Healthy infants and children as determined by medical history, physical examination, and judgment of the investigator.

Exclusion Criteria:

* Participation in other studies involving investigational drug(s)/vaccine(s) since birth (Cohort 1 only) or in the 6 months prior to study entry (Cohorts 2, 3, and 4) and/or during study participation.
* Other acute or chronic medical or psychiatric condition, including recent laboratory abnormality, that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Vaccination with licensed or investigational pneumococcal vaccine.
* Previous vaccination with licensed or investigational Hib vaccine.

Ages: 42 Days to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 936 (Actual)
Dates: Start 2018-06-23 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2023-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- China (2):
  - Huaiyin District Center for Disease Prevention and Control, Huaian, Jiangsu
  - Guanyun County Disease Control and Prevention, Lianyungang, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Chu K, Hu Y, Pan H, Wu J, Zhu D, Young MM Jr, Luo L, Yi Z, Giardina PC, Gruber WC, Scott DA, Watson W. A randomized, open-label, phase 3 study evaluating safety and immunogenicity of 13-valent pneumococcal conjugate vaccine in Chinese infants and children under 6 years of age. Hum Vaccin Immunother. 2023 Aug 1;19(2):2235926. doi: 10.1080/21645515.2023.2235926. PMID 37549923
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1851178

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study presents results following completion of all vaccinations, including data from 6-month follow-up after the last study vaccination. This study was conducted in China.
Pre-assignment Details: With the 280 additional participants included, a total of 986 participants were screened in this study, of whom 936 participants were enrolled or randomized, and 932 of 936 participants were vaccinated.
Groups:
- Cohort 1: Participants vaccinated 4 doses of 13vPnC (single intramuscular injection): Vaccination 1 (Visit 1): 42 to 56 days of age; Vaccination 2 (Visit 2): 42 to 70 days after Visit 1; Vaccination 3 (Visit 3): 42 to 70 days after Visit 2; Vaccination 4: 365 to 455 days of age.
- Cohort 2_13vPnC: Participants vaccinated 3 doses of 13vPnC (single intramuscular injection): Vaccination 1 (Visit 1): 7 to <12 months of age; Vaccination 2 (Visit 2): at least 28 days after Visit 1; Vaccination 3: 365 days to <450 days of age and at least 56 days after Visit 2.
- Cohort 2_Hib Vaccine: Participants vaccinated 2 doses of Hib Vaccine (single intramuscular injection): Vaccination 1 (Visit 1): 7 to <12 months of age; Vaccination 2: at least 28 days after Visit 1.
- Cohort 3_13vPnC: Participants vaccinated 2 doses of 13vPnC (single intramuscular injection): Vaccination 1 (Visit 1): >=1 to <2 years of age; Vaccination 2: at least 56 days after Visit 1.
- Cohort 3_Hib Vaccine: Participants vaccinated 1 dose of Hib vaccine (single intramuscular injection): Vaccination 1: >=1 to <2 years of age.
- Cohort 4_13vPnC: Participants vaccinated 1 dose of 13vPnC (single intramuscular injection): Vaccination 1: >=2 to <6 years of age.
- Cohort 4_Hib Vaccine: Participants vaccinated 1 dose of Hib vaccine (single intramuscular injection): Vaccination 1: >=2 to <6 years of age.
Period: Vaccination Period
Arm/Group | Cohort 1 | Cohort 2_13vPnC | Cohort 2_Hib Vaccine | Cohort 3_13vPnC | Cohort 3_Hib Vaccine | Cohort 4_13vPnC | Cohort 4_Hib Vaccine
Started | 125 | 236 | 117 | 165 | 83 | 138 | 68
Vaccination 1 | 125 | 236 | 117 | 165 | 83 | 138 | 68
Vaccination 2 | 114 | 219 | 107 | 146 | 0 | 0 | 0
Vaccination 3 | 111 | 214 | 0 | 0 | 0 | 0 | 0
Vaccination 4 | 92 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 90 | 214 | 107 | 146 | 83 | 138 | 68
Not Completed | 35 | 22 | 10 | 19 | 0 | 0 | 0
Not completed — Noncompliance With Investigational Product | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Parent/guardian | 26 | 21 | 10 | 19 | 0 | 0 | 0
Not completed — Other | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Follow-up Period
Arm/Group | Cohort 1 | Cohort 2_13vPnC | Cohort 2_Hib Vaccine | Cohort 3_13vPnC | Cohort 3_Hib Vaccine | Cohort 4_13vPnC | Cohort 4_Hib Vaccine
Started | 90 | 214 | 107 | 146 | 83 | 138 | 68
Completed | 89 | 201 | 98 | 137 | 76 | 131 | 67
Not Completed | 1 | 13 | 9 | 9 | 7 | 7 | 1
Not completed — Withdrawal by parent/guardian | 1 | 13 | 9 | 9 | 7 | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Participants vaccinated the first 3 of doses of 13vPnC (single intramuscular injection): Vaccination 1 (Visit 1): 42 to 56 days of age; Vaccination 2 (Visit 2): 42 to 70 days after Visit 1; Vaccination 3: 42 to 70 days after Visit 2; Vaccination 4: 365 to 455 days of age.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2_13vPnC | Cohort 2_Hib Vaccine | Cohort 3_13vPnC | Cohort 3_Hib Vaccine | Cohort 4_13vPnC | Cohort 4_Hib Vaccine | Total
Number analyzed (Participants) | 125 | 236 | 117 | 165 | 83 | 138 | 68 | 932
Age, Continuous [Mean (Standard Deviation); unit: Days] — Population: The ages of participants in Cohort 1 and 2 were counted in different 'Unit of Measures' from Cohort 3 and 4, and thus they were reported in separated 'Baseline Measures'. Cohort 1 and 2 were reported here.
  Days
    number analyzed (Participants) | 125 | 236 | 117 | 0 | 0 | 0 | 0 | 478
    (all) | 49.1 (3.78) | 286.0 (41.06) | 285.9 (40.40) |  |  |  |  | 224.0 (109.94)
Age, Continuous [Median (Full Range); unit: Days] — Population: The ages of participants in Cohort 1 and 2 were counted in different 'Unit of Measures' from Cohort 3 and 4, and thus they were reported in separated 'Baseline Measures'. Cohort 1 and 2 were reported here.
  Days
    number analyzed (Participants) | 125 | 236 | 117 | 0 | 0 | 0 | 0 | 478
    (all) | 49.0 [43 to 56] | 284.0 [216 to 361] | 281.0 [217 to 360] |  |  |  |  | 260.0 [43 to 361]
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The ages of participants in Cohort 1 and 2 were counted in different 'Unit of Measures' from Cohort 3 and 4, and thus they were reported in separated 'Baseline Measures'. Cohort 3 and 4 were reported here.
  Years
    number analyzed (Participants) | 0 | 0 | 0 | 165 | 83 | 138 | 68 | 454
    (all) |  |  |  | 1.5 (0.27) | 1.6 (0.30) | 3.3 (1.11) | 3.3 (1.04) | 2.3 (1.18)
Age, Continuous [Median (Full Range); unit: Years] — Population: The ages of participants in Cohort 1 and 2 were counted in different 'Unit of Measures' from Cohort 3 and 4, and thus they were reported in separated 'Baseline Measures'. Cohort 3 and 4 were reported here.
  Years
    number analyzed (Participants) | 0 | 0 | 0 | 165 | 83 | 138 | 68 | 454
    (all) |  |  |  | 1.5 [1 to 2] | 1.6 [1 to 2] | 3.1 [2 to 6] | 3.3 [2 to 6] | 1.9 [1 to 6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 115 | 50 | 83 | 36 | 56 | 37 | 436
  Male | 66 | 121 | 67 | 82 | 47 | 82 | 31 | 496
Race/Ethnicity, Customized [Number; unit: Participants]
  Race_Asian | 125 | 236 | 117 | 165 | 83 | 138 | 68 | 932
  Ethnicity_Non-Hispanic/Non-Latino | 125 | 236 | 117 | 165 | 83 | 138 | 68 | 932

OUTCOME MEASURES:

1. Primary Outcome: The Serotype-specific Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) for Each of the Pneumococcal Serotypes Measured in Cohorts 2, 3 and 4 Compared to IgG GMCs Measured in Cohort 1
Description: Serotype-specific IgG concentrations to the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in all participants from the blood samples taken 1 month after the infant series in Cohort 1 and the last dose 13vPnC in Cohorts 2, 3, 4. GMC and corresponding 2-sided 95% confidence intervals (CI) were evaluated. Geometric means (GMs) were calculated using all participants with available data for the specified blood draw.
Time Frame: Cohort 1: 1 month after the 3rd dose of 13vPnC (infant series dose). Cohort 2, 3, 4: 1 month after the last dose of 13vPnC.
Population: Evaluable analysis set included all participants evaluable for the study at randomization; received all study vaccinations for Cohort 2-4, received all 3 infant series doses for Cohort 1; had blood draw for assay testing within 27-56 days after 3rd vaccination for Cohort 1, visit 3 for Cohort 2, visit 2 for Cohort 3 and visit 1 for Cohort 4 and the sample from this blood draw provided at least 1 valid and determinate assay result; received no prohibited vaccine; had no major protocol violation.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Groups:
- Cohort 1_Infant Series: Participants vaccinated 3 infant series doses of 13vPnC (single intramuscular injection): Vaccination 1 (Visit 1): 42 to 56 days of age; Vaccination 2 (Visit 2): 42 to 70 days after Visit 1; Vaccination 3: 42 to 70 days after Visit 2.
- Cohort 4_vPnC: Participants vaccinated 1 dose of 13vPnC (single intramuscular injection): Vaccination 1: >=2 to <6 years of age.
Arm/Group | Cohort 1_Infant Series | Cohort 2_13vPnC | Cohort 3_13vPnC | Cohort 4_vPnC
Number analyzed (Participants) | 72 | 176 | 127 | 131
mcg/mL
  Serotype 1 | 5.40 [4.43 to 6.58] | 3.75 [3.26 to 4.32] | 4.38 [3.75 to 5.11] | 4.40 [3.76 to 5.14]
  Serotype 3 | 0.63 [0.54 to 0.75] | 1.19 [1.08 to 1.32] | 1.32 [1.16 to 1.51] | 1.12 [0.97 to 1.29]
  Serotype 4 | 3.96 [3.24 to 4.84] | 2.97 [2.60 to 3.40] | 4.04 [3.48 to 4.68] | 4.47 [3.92 to 5.10]
  Serotype 5 | 3.50 [2.91 to 4.19] | 3.07 [2.73 to 3.46] | 2.57 [2.26 to 2.92] | 2.92 [2.57 to 3.32]
  Serotype 6A | 5.35 [4.44 to 6.44] | 3.12 [2.74 to 3.57] | 3.19 [2.69 to 3.78] | 3.39 [2.80 to 4.09]
  Serotype 6B | 4.62 [3.76 to 5.69] | 2.20 [1.91 to 2.54] | 2.47 [2.06 to 2.96] | 2.96 [2.44 to 3.59]
  Serotype 7F | 7.14 [6.00 to 8.50] | 5.73 [5.10 to 6.44] | 7.87 [6.90 to 8.96] | 7.08 [6.19 to 8.10]
  Serotype 9V | 3.66 [2.99 to 4.50] | 2.24 [1.99 to 2.51] | 3.31 [2.90 to 3.77] | 3.68 [3.22 to 4.21]
  Serotype 14 | 15.09 [11.39 to 20.00] | 10.89 [9.59 to 12.35] | 9.79 [8.40 to 11.41] | 6.94 [5.53 to 8.70]
  Serotype 18C | 4.94 [4.11 to 5.94] | 2.25 [1.98 to 2.57] | 3.88 [3.25 to 4.64] | 5.60 [4.74 to 6.62]
  Serotype 19A | 3.44 [2.85 to 4.16] | 3.62 [3.30 to 3.97] | 5.55 [4.86 to 6.34] | 11.62 [9.75 to 13.86]
  Serotype 19F | 4.95 [3.91 to 6.26] | 4.50 [3.98 to 5.09] | 5.04 [4.28 to 5.92] | 5.44 [4.46 to 6.64]
  Serotype 23F | 4.36 [3.23 to 5.88] | 2.04 [1.76 to 2.37] | 2.26 [1.90 to 2.67] | 2.80 [2.33 to 3.36]

2. Primary Outcome: Number of Participants With Local Reactions and Systemic Events Within 7 Days After Each Vaccination in Cohort 2
Description: Local reactions (redness, swelling, and tenderness) at the site of the investigational product injection were monitored daily for 7 days after each vaccination. Temperature were collected at bedtime daily for 7 days and at any time during the 7 days that fever is suspected. Fever is defined as temperature of greater than or equal to 38.0ºC (100.4ºF). Other systemic events (decreased appetite, drowsiness and irritability) were recorded for 7 days after each investigational product vaccination.
Time Frame: Within 7 Days After Each Vaccination
Population: The safety population included all participants who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2_13vPnC_Vaccination 1; Cohort 2_13vPnC_Vaccination 2; Cohort 2_13vPnC_Vaccination 3: Participants vaccinated 3 doses of 13vPnC (single intramuscular injection): Vaccination 1 (Visit 1): 7 to <12 months of age; Vaccination 2 (Visit 2): at least 28 days after Visit 1; Vaccination 3: 365 days to <450 days of age and at least 56 days after Visit 2.
- Cohort 2_Hib Vaccine_Vaccination 1; Cohort 2_Hib Vaccine_Vaccination 2: Participants vaccinated 2 doses of Hib Vaccine (single intramuscular injection): Vaccination 1 (Visit 1): 7 to <12 months of age; Vaccination 2: at least 28 days after Visit 1.
Arm/Group | Cohort 2_13vPnC_Vaccination 1 | Cohort 2_Hib Vaccine_Vaccination 1 | Cohort 2_13vPnC_Vaccination 2 | Cohort 2_Hib Vaccine_Vaccination 2 | Cohort 2_13vPnC_Vaccination 3
Number analyzed (Participants) | 236 | 117 | 219 | 107 | 194
Participants
  Local Reactions | 66 | 18 | 20 | 14 | 4
  Systemic Events | 23 | 7 | 23 | 5 | 1

3. Primary Outcome: Number of Participants With Local Reactions and Systemic Events Within 7 Days After Each Vaccination in Cohort 3
Description: as for outcome 2
Time Frame: Within 7 Days After Each Vaccination
Population: The safety population included all participants who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 3_13vPnC _Vaccination 1; Cohort 3_13vPnC _Vaccination 2: Participants vaccinated 2 doses of 13vPnC (single intramuscular injection): Vaccination 1 (Visit 1): >=1 to <2 years of age; Vaccination 2: at least 56 days after Visit 1.
- Cohort 3_Hib Vaccine_Vaccination 1: Participants vaccinated 1 dose of Hib vaccine (single intramuscular injection): Vaccination 1: >=1 to <2 years of age; Participant did not receive Hib vaccine at Visit 2.
Arm/Group | Cohort 3_13vPnC _Vaccination 1 | Cohort 3_Hib Vaccine_Vaccination 1 | Cohort 3_13vPnC _Vaccination 2
Number analyzed (Participants) | 164 | 83 | 146
Participants
  Local Reactions | 45 | 10 | 9
  Systemic Events | 26 | 7 | 4

4. Primary Outcome: Number of Participants With Local Reactions and Systemic Events Within 7 Days After Each Vaccination in Cohort 4
Description: Local reactions (redness, swelling, and tenderness) at the site of the investigational product injection were monitored daily for 7 days after each vaccination. Temperature were collected at bedtime daily for 7 days and at any time during the 7 days that fever is suspected. Fever is defined as temperature of greater than or equal to 38.0ºC (100.4ºF). Other systemic events (fatigue, headache, vomiting, diarrhea, muscle pain and joint pain) were recorded for 7 days after each investigational product vaccination.
Time Frame: Within 7 Days After Each Vaccination
Population: The safety population included all participants who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 4_13vPnC_Vaccination 1: Participants vaccinated 1 dose of 13vPnC (single intramuscular injection): Vaccination 1: >=2 to <6 years of age.
- Cohort 4_Hib Vaccine_Vaccination 1: Participants vaccinated 1 dose of Hib vaccine (single intramuscular injection): Vaccination 1: >=2 to <6 years of age.
Arm/Group | Cohort 4_13vPnC_Vaccination 1 | Cohort 4_Hib Vaccine_Vaccination 1
Number analyzed (Participants) | 138 | 68
Participants
  Local Reactions: number analyzed (Participants) | 138 | 67
  Local Reactions | 48 | 21
  Systemic Events | 17 | 10

5. Primary Outcome: Number of Participants With Adverse Event (AE) From the Signing of the Informed Consent Document (ICD) to 1 Month After the Last Vaccination in Cohorts 2, 3, 4
Description: An AE was any untoward medical occurrence in a study participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage.
Time Frame: From the signing of ICD to 1 month after the last vaccination (13vPnC or Hib) in Cohort 2, 3 and 4.
Population: The safety population included all participants who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 3_Hib Vaccine: Participants vaccinated 1 dose of Hib vaccine (single intramuscular injection): Vaccination 1: >=1 to <2 years of age; Participant did not receive Hib vaccine at Visit 2.
Arm/Group | Cohort 2_13vPnC | Cohort 2_Hib Vaccine | Cohort 3_13vPnC | Cohort 3_Hib Vaccine | Cohort 4_13vPnC | Cohort 4_Hib Vaccine
Number analyzed (Participants) | 236 | 117 | 165 | 83 | 138 | 68
Participants | 76 | 29 | 21 | 1 | 11 | 1

6. Primary Outcome: Number of Participants With Newly Diagnosed Chronic Medical Conditions (NDCMCs) From 1 Month to 6 Months After the Last Vaccination in Cohorts 2, 3, 4
Description: Number of participants with NDCMCs from 1 month after the last study vaccination (13vPnC or Hib vaccine) to 6 months after the last study vaccination in Cohorts 2, 3, and 4. An NDCMC was defined as a disease or medical condition that was not identified prior to study start and was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: From 1 month to 6 months (5 months) after the last vaccination in Cohorts 2,3,4.
Population: The safety population included all participants who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2_Hib Vaccine: Participants vaccinated 2 doses of Hib Vaccine (single intramuscular injection): Vaccination 1 (Visit 1): 7 to <12 months of age; Vaccination 2 (Visit 2): at least 28 days after Visit 1.
Arm/Group | Cohort 2_13vPnC | Cohort 2_Hib Vaccine | Cohort 3_13vPnC | Cohort 3_Hib Vaccine | Cohort 4_13vPnC | Cohort 4_Hib Vaccine
Number analyzed (Participants) | 236 | 117 | 165 | 83 | 138 | 68
Participants | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With SAE From the Signing of the ICD to 6 Months After the Last Vaccination in Cohorts 2, 3, 4
Description: An SAE was any untoward medical occurrence at any dose that resulted in death, was life-threatening (immediate risk of death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect or considered to be an important medical event.
Time Frame: From the signing of ICD to 6 month after the last vaccination (13vPnC or Hib) in Cohorts 2, 3 and 4.
Population: The safety population included all participants who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2_13vPnC | Cohort 2_Hib Vaccine | Cohort 3_13vPnC | Cohort 3_Hib Vaccine | Cohort 4_13vPnC | Cohort 4_Hib Vaccine
Number analyzed (Participants) | 236 | 117 | 165 | 83 | 138 | 68
Participants | 5 | 1 | 2 | 0 | 2 | 1

8. Secondary Outcome: The Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) for Each of the Pneumococcal Serotypes Measured in Cohorts 2, 3 and 4 Compared to IgG GMTs Measured in Cohort 1.
Description: Serotype-specific OPA titers to the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in a randomly selected subset of about 50 participants receiving 13vPnC from the blood samples taken 1 month after the infant series in Cohort 1 and the last 13vPnC vaccination in each of the 3 cohorts. GMT and corresponding 2-sided 95% CI were evaluated. GMs were calculated using all participants with available data for the specified blood draw.
Time Frame: Cohort 1: 1 month after the 3rd dose of 13vPnC. Cohort 2, 3, 4: 1 month after the last dose of 13vPnC.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Groups:
- Cohort 1_Infant Series: Participants vaccinated 3 infant series doses of 13vPnC (single intramuscular injection): Vaccination 1: 42 to 56 days of age; Vaccination 2: 42 to 70 days after Visit 1; Vaccination 3: 42 to 70 days after Visit 2.
- Cohort 2_13vPnC: Participants vaccinated 3 doses of 13vPnC (single intramuscular injection): Vaccination 1: 7 to <12 months of age; Vaccination 2: at least 28 days after Visit 1; Vaccination 3: 365 days to <450 days of age and at least 56 days after Visit 2.
- Cohort 3_13vPnC: Participants vaccinated 2 doses of 13vPnC (single intramuscular injection): Vaccination 1: >=1 to <2 years of age; Vaccination 2: at least 56 days after Visit 1.
Arm/Group | Cohort 1_Infant Series | Cohort 2_13vPnC | Cohort 3_13vPnC | Cohort 4_13vPnC
Number analyzed (Participants) | 37 | 87 | 78 | 71
GMT
  Serotype 1 | 201.7 [134.8 to 301.8] | 142.7 [103.4 to 196.9] | 93.3 [70.1 to 124.1] | 40.9 [31.3 to 53.4]
  Serotype 3 | 112.9 [82.5 to 154.4] | 249.0 [205.7 to 301.5] | 332.3 [273.3 to 404.1] | 244.8 [192.0 to 312.1]
  Serotype 4 | 1857.8 [1264.8 to 2728.8] | 2172.2 [1740.7 to 2710.7] | 2682.8 [2210.4 to 3256.2] | 4236.3 [3489.6 to 5142.8]
  Serotype 5 | 645.9 [452.6 to 921.8] | 286.3 [214.5 to 382.0] | 164.5 [131.5 to 205.7] | 79.3 [57.7 to 109.0]
  Serotype 6A | 5996.2 [4337.5 to 8289.3] | 6042.7 [4830.2 to 7559.6] | 7661.8 [6116.0 to 9598.4] | 5849.3 [4364.0 to 7840.2]
  Serotype 6B | 2331.6 [1481.3 to 3670.0] | 2181.6 [1350.1 to 3525.2] | 4986.3 [3717.6 to 6687.9] | 3775.2 [2825.1 to 5044.9]
  Serotype 7F | 10413.4 [7373.1 to 14707.3] | 10234.6 [8612.2 to 12162.8] | 14963.5 [12367.6 to 18104.4] | 17107.3 [13842.7 to 21141.8]
  Serotype 9V | 5386.5 [3634.0 to 7984.3] | 4154.1 [3358.6 to 5138.0] | 7220.1 [5620.9 to 9274.2] | 10533.5 [7811.9 to 14203.4]
  Serotype 14 | 2859.4 [1688.9 to 4899.3] | 4108.0 [3342.6 to 5048.8] | 6885.4 [5642.6 to 8402.0] | 7504.5 [5718.2 to 9848.9]
  Serotype 18C | 2677.9 [2000.3 to 3585.0] | 1486.6 [1124.6 to 1965.2] | 1890.4 [1429.0 to 2500.6] | 2111.9 [1630.6 to 2735.2]
  Serotype 19A | 1677.3 [1159.9 to 2425.5] | 2611.3 [2071.6 to 3291.6] | 3560.0 [2867.8 to 4419.1] | 3055.1 [2154.1 to 4333.1]
  Serotype 19F | 744.4 [506.7 to 1093.6] | 1158.4 [937.0 to 1432.1] | 1854.0 [1520.3 to 2260.8] | 1629.7 [1292.9 to 2054.2]
  Serotype 23F | 3833.2 [2216.2 to 6630.1] | 5640.0 [3590.5 to 8859.4] | 6693.6 [4464.2 to 10036.4] | 4234.7 [2916.1 to 6149.5]

9. Secondary Outcome: The Serotype-specific IgG GMCs for Each of the Pneumococcal Serotypes in Cohorts 2, 3, 4 Vaccinated With 13 vPnC Compared to Cohorts 2, 3 and 4 Vaccinated With Hib Vaccine.
Description: Serotype-specific IgG concentrations to the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in all participants from the blood samples taken before vaccination and 1 month after vaccination in each of the 3 cohorts. GMC and corresponding 2-sided 95% CI were evaluated. GMs were calculated using all participants with available data for the specified blood draw.
Time Frame: Cohort 2, 3, 4: Before Vaccination and 1 Month After the Last Dose
Population: Evaluable analysis set included all participants evaluable for the study at randomization; received all study vaccinations for Cohort 2-4; had blood draw for assay testing within 27-56 days after visit 3 for Cohort 2, visit 2 for Cohort 3 and visit 1 for Cohort 4 and the sample from this blood draw provided at least 1 valid and determinate assay result; received no prohibited vaccine; had no major protocol violation.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Groups:
- Cohort 2_Hib Vaccine: Participants vaccinated 2 doses of Hib Vaccine (single intramuscular injection): Vaccination 1: 7 to <12 months of age; Vaccination 2: at least 28 days after Visit 1.
Arm/Group | Cohort 2_13vPnC | Cohort 2_Hib Vaccine | Cohort 3_13vPnC | Cohort 3_Hib Vaccine | Cohort 4_13vPnC | Cohort 4_Hib Vaccine
Number analyzed (Participants) | 176 | 72 | 127 | 77 | 131 | 67
mcg/mL
  Serotype 1 - Before Vaccination: number analyzed (Participants) | 176 | 72 | 126 | 77 | 131 | 67
  Serotype 1 - Before Vaccination | 0.02 [0.01 to 0.02] | 0.02 [0.01 to 0.03] | 0.07 [0.05 to 0.09] | 0.07 [0.05 to 0.10] | 0.18 [0.14 to 0.22] | 0.21 [0.15 to 0.28]
  Serotype 1 - 1 Month After the Last Dose | 3.75 [3.26 to 4.32] | 0.04 [0.03 to 0.06] | 4.38 [3.75 to 5.11] | 0.07 [0.04 to 0.11] | 4.40 [3.76 to 5.14] | 0.16 [0.12 to 0.23]
  Serotype 3 - Before Vaccination: number analyzed (Participants) | 176 | 72 | 125 | 77 | 131 | 67
  Serotype 3 - Before Vaccination | 0.03 [0.03 to 0.04] | 0.03 [0.02 to 0.04] | 0.07 [0.05 to 0.09] | 0.07 [0.05 to 0.09] | 0.14 [0.10 to 0.18] | 0.13 [0.08 to 0.22]
  Serotype 3 - 1 Month After the Last Dose | 1.19 [1.08 to 1.32] | 0.04 [0.03 to 0.05] | 1.32 [1.16 to 1.51] | 0.09 [0.06 to 0.13] | 1.12 [0.97 to 1.29] | 0.12 [0.07 to 0.20]
  Serotype 4 - Before Vaccination | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.01] | 0.03 [0.02 to 0.04] | 0.04 [0.03 to 0.06] | 0.07 [0.05 to 0.10] | 0.07 [0.05 to 0.11]
  Serotype 4 - 1 Month After the Last Dose | 2.97 [2.60 to 3.40] | 0.02 [0.01 to 0.02] | 4.04 [3.48 to 4.68] | 0.03 [0.02 to 0.05] | 4.47 [3.92 to 5.10] | 0.06 [0.04 to 0.08]
  Serotype 5 - Before Vaccination | 0.38 [0.34 to 0.43] | 0.36 [0.31 to 0.42] | 0.69 [0.60 to 0.78] | 0.63 [0.54 to 0.74] | 1.04 [0.92 to 1.17] | 0.97 [0.83 to 1.13]
  Serotype 5 - 1 Month After the Last Dose | 3.07 [2.73 to 3.46] | 0.51 [0.43 to 0.61] | 2.57 [2.26 to 2.92] | 0.74 [0.62 to 0.88] | 2.92 [2.57 to 3.32] | 0.89 [0.73 to 1.07]
  Serotype 6A - Before Vaccination: number analyzed (Participants) | 174 | 72 | 127 | 76 | 129 | 67
  Serotype 6A - Before Vaccination | 0.15 [0.13 to 0.18] | 0.16 [0.13 to 0.20] | 0.30 [0.26 to 0.35] | 0.36 [0.30 to 0.42] | 0.79 [0.68 to 0.93] | 0.79 [0.64 to 0.97]
  Serotype 6A - 1 Month After the Last Dose: number analyzed (Participants) | 176 | 72 | 127 | 77 | 129 | 67
  Serotype 6A - 1 Month After the Last Dose | 3.12 [2.74 to 3.57] | 0.20 [0.15 to 0.26] | 3.19 [2.69 to 3.78] | 0.42 [0.34 to 0.51] | 3.39 [2.80 to 4.09] | 0.80 [0.65 to 0.98]
  Serotype 6B - Before Vaccination | 0.15 [0.12 to 0.17] | 0.15 [0.11 to 0.19] | 0.30 [0.26 to 0.35] | 0.35 [0.30 to 0.41] | 0.80 [0.69 to 0.94] | 0.70 [0.58 to 0.84]
  Serotype 6B - 1 Month After the Last Dose | 2.20 [1.91 to 2.54] | 0.21 [0.16 to 0.26] | 2.47 [2.06 to 2.96] | 0.38 [0.32 to 0.46] | 2.96 [2.44 to 3.59] | 0.62 [0.49 to 0.79]
  Serotype 7F - Before Vaccination: number analyzed (Participants) | 175 | 72 | 127 | 76 | 130 | 64
  Serotype 7F - Before Vaccination | 0.03 [0.03 to 0.04] | 0.03 [0.02 to 0.04] | 0.10 [0.08 to 0.12] | 0.11 [0.08 to 0.15] | 0.25 [0.21 to 0.31] | 0.25 [0.18 to 0.33]
  Serotype 7F - 1 Month After the Last Dose: number analyzed (Participants) | 176 | 71 | 127 | 76 | 131 | 67
  Serotype 7F - 1 Month After the Last Dose | 5.73 [5.10 to 6.44] | 0.05 [0.03 to 0.07] | 7.87 [6.90 to 8.96] | 0.13 [0.09 to 0.20] | 7.08 [6.19 to 8.10] | 0.21 [0.16 to 0.29]
  Serotype 9V - Before Vaccination: number analyzed (Participants) | 176 | 72 | 126 | 77 | 131 | 67
  Serotype 9V - Before Vaccination | 0.13 [0.11 to 0.16] | 0.16 [0.12 to 0.22] | 0.25 [0.20 to 0.31] | 0.27 [0.23 to 0.33] | 0.55 [0.47 to 0.65] | 0.41 [0.31 to 0.55]
  Serotype 9V - 1 Month After the Last Dose: number analyzed (Participants) | 176 | 72 | 127 | 76 | 131 | 67
  Serotype 9V - 1 Month After the Last Dose | 2.24 [1.99 to 2.51] | 0.20 [0.14 to 0.27] | 3.31 [2.90 to 3.77] | 0.34 [0.26 to 0.43] | 3.68 [3.22 to 4.21] | 0.45 [0.37 to 0.54]
  Serotype 14 - Before Vaccination: number analyzed (Participants) | 175 | 72 | 127 | 77 | 130 | 67
  Serotype 14 - Before Vaccination | 0.03 [0.02 to 0.04] | 0.02 [0.02 to 0.03] | 0.03 [0.03 to 0.05] | 0.05 [0.03 to 0.09] | 0.19 [0.12 to 0.29] | 0.20 [0.11 to 0.36]
  Serotype 14 - 1 Month After the Last Dose | 10.89 [9.59 to 12.35] | 0.02 [0.02 to 0.03] | 9.79 [8.40 to 11.41] | 0.07 [0.04 to 0.11] | 6.94 [5.53 to 8.70] | 0.20 [0.11 to 0.36]
  Serotype 18C - Before Vaccination: number analyzed (Participants) | 176 | 72 | 127 | 77 | 130 | 67
  Serotype 18C - Before Vaccination | 0.01 [0.01 to 0.01] | 0.01 [0.01 to 0.02] | 0.04 [0.03 to 0.06] | 0.05 [0.04 to 0.08] | 0.20 [0.15 to 0.27] | 0.20 [0.12 to 0.29]
  Serotype 18C - 1 Month After the Last Dose: number analyzed (Participants) | 176 | 72 | 127 | 77 | 131 | 66
  Serotype 18C - 1 Month After the Last Dose | 2.25 [1.98 to 2.57] | 0.02 [0.01 to 0.03] | 3.88 [3.25 to 4.64] | 0.07 [0.04 to 0.12] | 5.60 [4.74 to 6.62] | 0.18 [0.11 to 0.29]
  Serotype 19A - Before Vaccination | 0.36 [0.31 to 0.41] | 0.38 [0.31 to 0.46] | 0.65 [0.55 to 0.76] | 0.69 [0.58 to 0.83] | 1.72 [1.46 to 2.02] | 1.44 [1.13 to 1.83]
  Serotype 19A - 1 Month After the Last Dose | 3.62 [3.30 to 3.97] | 0.50 [0.41 to 0.60] | 5.55 [4.86 to 6.34] | 0.88 [0.71 to 1.10] | 11.62 [9.75 to 13.86] | 1.33 [1.04 to 1.70]
  Serotype 19F - Before Vaccination: number analyzed (Participants) | 173 | 72 | 127 | 77 | 131 | 67
  Serotype 19F - Before Vaccination | 0.08 [0.07 to 0.11] | 0.11 [0.08 to 0.16] | 0.23 [0.18 to 0.29] | 0.23 [0.17 to 0.31] | 0.62 [0.49 to 0.78] | 0.57 [0.41 to 0.80]
  Serotype 19F - 1 Month After the Last Dose | 4.50 [3.98 to 5.09] | 0.13 [0.09 to 0.19] | 5.04 [4.28 to 5.92] | 0.27 [0.18 to 0.39] | 5.44 [4.46 to 6.64] | 0.53 [0.38 to 0.73]
  Serotype 23F - Before Vaccination: number analyzed (Participants) | 176 | 72 | 126 | 76 | 131 | 67
  Serotype 23F - Before Vaccination | 0.11 [0.10 to 0.13] | 0.11 [0.09 to 0.14] | 0.19 [0.17 to 0.23] | 0.22 [0.19 to 0.26] | 0.54 [0.46 to 0.64] | 0.45 [0.35 to 0.57]
  Serotype 23F - 1 Month After the Last Dose: number analyzed (Participants) | 176 | 71 | 127 | 77 | 131 | 67
  Serotype 23F - 1 Month After the Last Dose | 2.04 [1.76 to 2.37] | 0.17 [0.14 to 0.21] | 2.26 [1.90 to 2.67] | 0.27 [0.22 to 0.34] | 2.80 [2.33 to 3.36] | 0.44 [0.34 to 0.56]

10. Secondary Outcome: The Serotype-specific OPA GMT for Each of the Pneumococcal Serotypes in Cohorts 2, 3, 4 Vaccinated With 13 vPnC Compared to Cohorts 2, 3 and 4 Vaccinated With Hib Vaccine.
Description: Serotype-specific OPA titers to the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in a randomly selected subset of approximately 50 participants receiving 13vPnC and approximately 25 participants receiving Hib vaccine from the blood samples taken before vaccination and 1 month after the last 13vPnC vaccination in each of the 3 cohorts.
Time Frame: Cohort 2, 3, 4: Before Vaccination and 1 Month After the Last Dose
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | Cohort 2_13vPnC | Cohort 2_Hib Vaccine | Cohort 3_13vPnC | Cohort 3_Hib Vaccine | Cohort 4_13vPnC | Cohort 4_Hib Vaccine
Number analyzed (Participants) | 87 | 34 | 78 | 42 | 71 | 36
GMT
  Serotype 1 - Before Vaccination | 4.1 [3.9 to 4.4] | 4.2 [3.8 to 4.6] | 4.0 [4.0 to 4.0] | 4.2 [3.8 to 4.7] | 4.6 [4.2 to 5.0] | 5.5 [4.5 to 6.7]
  Serotype 1 - 1 Month After the Last Dose | 142.7 [103.4 to 196.9] | 4.9 [3.6 to 6.8] | 93.3 [70.1 to 124.1] | 4.8 [3.8 to 6.0] | 40.9 [31.3 to 53.4] | 4.4 [3.8 to 5.1]
  Serotype 3 - Before Vaccination | 5.8 [5.0 to 6.7] | 6.7 [4.5 to 10.0] | 11.9 [8.6 to 16.5] | 11.3 [6.9 to 18.5] | 27.1 [19.2 to 38.4] | 40.0 [22.7 to 70.7]
  Serotype 3 - 1 Month After the Last Dose | 249.0 [205.7 to 301.5] | 7.4 [4.9 to 11.3] | 332.3 [273.3 to 404.1] | 13.4 [7.7 to 23.4] | 244.8 [192.0 to 312.1] | 28.4 [16.2 to 49.7]
  Serotype 4 - Before Vaccination | 5.5 [4.3 to 6.9] | 5.0 [3.6 to 6.9] | 6.3 [4.8 to 8.3] | 9.5 [5.6 to 16.2] | 23.4 [13.8 to 39.7] | 15.9 [8.4 to 30.1]
  Serotype 4 - 1 Month After the Last Dose | 2172.2 [1740.7 to 2710.7] | 10.3 [5.2 to 20.3] | 2682.8 [2210.4 to 3256.2] | 10.6 [5.7 to 19.6] | 4236.3 [3489.6 to 5142.8] | 19.2 [10.0 to 36.6]
  Serotype 5 - Before Vaccination | 4.3 [3.8 to 4.9] | 4.0 [4.0 to 4.0] | 4.2 [3.9 to 4.4] | 4.1 [3.9 to 4.4] | 4.7 [4.1 to 5.3] | 4.2 [3.9 to 4.6]
  Serotype 5 - 1 Month After the Last Dose | 286.3 [214.5 to 382.0] | 6.2 [4.0 to 9.7] | 164.5 [131.5 to 205.7] | 5.1 [3.6 to 7.2] | 79.3 [57.7 to 109.0] | 4.8 [4.0 to 5.8]
  Serotype 6A - Before Vaccination | 5.0 [4.1 to 6.3] | 4.0 [4.0 to 4.0] | 6.9 [4.9 to 9.8] | 8.2 [4.7 to 14.3] | 45.5 [26.5 to 78.0] | 137.4 [63.3 to 297.9]
  Serotype 6A - 1 Month After the Last Dose | 6042.7 [4830.2 to 7559.6] | 5.9 [4.0 to 8.8] | 7661.8 [6116.0 to 9598.4] | 17.8 [8.1 to 39.1] | 5849.3 [4364.0 to 7840.2] | 101.8 [45.7 to 226.8]
  Serotype 6B - Before Vaccination | 5.1 [4.1 to 6.4] | 4.0 [4.0 to 4.0] | 8.2 [5.5 to 12.2] | 9.7 [5.6 to 16.8] | 53.6 [30.4 to 94.5] | 94.9 [43.0 to 209.3]
  Serotype 6B - 1 Month After the Last Dose | 2181.6 [1350.1 to 3525.2] | 5.7 [3.8 to 8.6] | 4986.3 [3717.6 to 6687.9] | 20.2 [9.3 to 43.8] | 3775.2 [2825.1 to 5044.9] | 117.7 [51.9 to 267.1]
  Serotype 7F - Before Vaccination | 63.0 [35.8 to 111.0] | 29.6 [12.4 to 70.4] | 195.8 [114.5 to 334.9] | 432.7 [213.8 to 875.8] | 1155.2 [852.6 to 1565.2] | 892.7 [515.3 to 1546.5]
  Serotype 7F - 1 Month After the Last Dose | 10234.6 [8612.2 to 12162.8] | 94.0 [37.2 to 237.3] | 14963.5 [12367.6 to 18104.4] | 707.1 [361.9 to 1381.6] | 17107.3 [13842.7 to 21141.8] | 1090.7 [696.2 to 1708.8]
  Serotype 9V - Before Vaccination | 9.3 [6.3 to 13.8] | 11.3 [5.9 to 21.5] | 59.5 [34.1 to 103.7] | 74.5 [31.0 to 179.0] | 458.9 [280.9 to 749.8] | 850.2 [469.4 to 1539.9]
  Serotype 9V - 1 Month After the Last Dose | 4154.1 [3358.6 to 5138.0] | 20.6 [9.1 to 46.8] | 7220.1 [5620.9 to 9274.2] | 154.3 [69.9 to 340.9] | 10533.5 [7811.9 to 14203.4] | 795.1 [472.6 to 1337.6]
  Serotype 14 - Before Vaccination | 9.8 [6.5 to 14.7] | 12.7 [6.2 to 26.3] | 30.0 [16.1 to 56.1] | 19.1 [8.5 to 43.0] | 132.6 [64.8 to 271.5] | 210.6 [87.7 to 505.5]
  Serotype 14 - 1 Month After the Last Dose | 4108.0 [3342.6 to 5048.8] | 26.6 [11.4 to 62.3] | 6885.4 [5642.6 to 8402.0] | 39.0 [16.3 to 93.2] | 7504.5 [5718.2 to 9848.9] | 294.9 [126.5 to 687.1]
  Serotype 18C - Before Vaccination | 4.3 [3.8 to 4.9] | 4.4 [3.8 to 5.1] | 6.1 [5.0 to 7.4] | 6.3 [4.4 to 8.9] | 12.7 [8.4 to 19.1] | 20.3 [10.0 to 41.3]
  Serotype 18C - 1 Month After the Last Dose | 1486.6 [1124.6 to 1965.2] | 6.5 [4.1 to 10.3] | 1890.4 [1429.0 to 2500.6] | 7.9 [4.8 to 13.1] | 2111.9 [1630.6 to 2735.2] | 24.6 [12.1 to 50.1]
  Serotype 19A - Before Vaccination | 5.3 [4.5 to 6.3] | 5.8 [4.1 to 8.1] | 11.1 [7.8 to 15.8] | 13.8 [7.8 to 24.3] | 60.3 [37.6 to 96.7] | 52.0 [24.2 to 111.6]
  Serotype 19A - 1 Month After the Last Dose | 2611.3 [2071.6 to 3291.6] | 6.4 [4.6 to 8.9] | 3560.0 [2867.8 to 4419.1] | 15.5 [8.6 to 28.2] | 3055.1 [2154.1 to 4333.1] | 54.3 [27.6 to 107.1]
  Serotype 19F - Before Vaccination | 4.3 [3.9 to 4.8] | 4.6 [3.7 to 5.7] | 6.2 [4.9 to 7.8] | 6.1 [4.5 to 8.3] | 24.7 [15.7 to 38.9] | 38.5 [18.1 to 81.8]
  Serotype 19F - 1 Month After the Last Dose | 1158.4 [937.0 to 1432.1] | 5.9 [4.1 to 8.6] | 1854.0 [1520.3 to 2260.8] | 9.5 [5.6 to 16.2] | 1629.7 [1292.9 to 2054.2] | 41.1 [19.4 to 86.8]
  Serotype 23F - Before Vaccination | 5.1 [4.1 to 6.3] | 4.7 [3.4 to 6.4] | 15.0 [8.8 to 25.6] | 11.1 [5.6 to 22.0] | 106.0 [59.5 to 188.9] | 70.5 [29.5 to 168.3]
  Serotype 23F - 1 Month After the Last Dose | 5640.0 [3950.5 to 8859.4] | 20.2 [8.5 to 47.7] | 6693.6 [4464.2 to 10036.4] | 19.4 [8.8 to 42.8] | 4234.7 [2916.1 to 6149.5] | 97.2 [40.8 to 231.2]

11. Secondary Outcome: Percentage of Participants Achieving Pneumococcal Serotype-specific IgG Concentration ≥0.35 mcg/mL for 1 Month After the Last Vaccination in Cohorts 2,3,4 (13vPnC and Hib Vaccine) and 1 Month After the Infant Series in Cohort 1 (13vPnC).
Description: Serotype-specific IgG concentrations to the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in all participants from the blood samples taken 1 month after the infant series in Cohort 1 and the last dose of vaccination (13vPnC or Hib vaccine) in Cohorts 2, 3, 4.
Time Frame: Cohort 1: 1 month after the 3rd dose of 13vPnC. Cohorts 2, 3, 4: 1 month after the last dose of 13vPnC and Hib Vaccine.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Cohort 1_Infant Series: Proportion of participants achieving pneumococcal serotype-specific IgG concentration >=0.35 µg/mL for 1 month after infant series in Cohort 1.
- Cohort 2_13vPnC: Proportion of participants achieving pneumococcal serotype-specific IgG concentration >=0.35 µg/mL for 1 month after the last dose of 13vPnC in Cohort 2.
- Cohort 2_Hib Vaccine: Proportion of participants achieving pneumococcal serotype-specific IgG concentration >=0.35 µg/mL for 1 month after the last dose of Hib vaccine in Cohort 2.
- Cohort 3_13vPnC: Proportion of participants achieving pneumococcal serotype-specific IgG concentration >=0.35 µg/mL for 1 month after the last dose of 13vPnC in Cohort 3.
- Cohort 3_Hib Vaccine: Proportion of participants achieving pneumococcal serotype-specific IgG concentration >=0.35 µg/mL for 1 month after the last dose of Hib vaccine in Cohort 3.
- Cohort 4_13vPnC: Proportion of participants achieving pneumococcal serotype-specific IgG concentration >=0.35 µg/mL for 1 month after the last dose of 13vPnC in Cohort 4.
- Cohort 4_Hib Vaccine: Proportion of participants achieving pneumococcal serotype-specific IgG concentration >=0.35 µg/mL for 1 month after the last dose of Hib vaccine in Cohort 4.
Arm/Group | Cohort 1_Infant Series | Cohort 2_13vPnC | Cohort 2_Hib Vaccine | Cohort 3_13vPnC | Cohort 3_Hib Vaccine | Cohort 4_13vPnC | Cohort 4_Hib Vaccine
Number analyzed (Participants) | 72 | 176 | 72 | 127 | 77 | 131 | 67
Percentage of Participants
  Serotype 1 | 100.0 [95.0 to 100.0] | 99.4 [96.9 to 100.0] | 4.2 [0.9 to 11.7] | 97.6 [93.3 to 99.5] | 10.4 [4.6 to 19.4] | 99.2 [95.8 to 100.0] | 23.9 [14.3 to 35.9]
  Serotype 3 | 83.3 [72.7 to 91.1] | 97.7 [94.3 to 99.4] | 4.2 [0.9 to 11.7] | 94.5 [89.0 to 97.8] | 11.7 [5.5 to 21.0] | 98.5 [94.6 to 99.8] | 19.4 [10.8 to 30.9]
  Serotype 4 | 100.0 [95.0 to 100.0] | 99.4 [96.9 to 100.0] | 5.6 [1.5 to 13.6] | 97.6 [93.3 to 99.5] | 6.5 [2.1 to 14.5] | 99.2 [95.8 to 100.0] | 4.5 [0.9 to 12.5]
  Serotype 5 | 100.0 [95.0 to 100.0] | 100.0 [97.9 to 100.0] | 69.4 [57.5 to 79.8] | 100.0 [97.1 to 100.0] | 85.7 [75.9 to 92.6] | 99.2 [95.8 to 100.0] | 88.1 [77.8 to 94.7]
  Serotype 6A: number analyzed (Participants) | 72 | 176 | 72 | 127 | 76 | 129 | 67
  Serotype 6A | 100.0 [95.0 to 100.0] | 97.7 [94.3 to 99.4] | 33.3 [22.7 to 45.4] | 97.6 [93.3 to 99.5] | 56.6 [44.7 to 67.9] | 100.0 [97.2 to 100.0] | 86.6 [76.0 to 93.7]
  Serotype 6B | 100.0 [95.0 to 100.0] | 96.0 [92.0 to 98.4] | 23.6 [14.4 to 35.1] | 97.6 [93.3 to 99.5] | 50.6 [39.0 to 62.2] | 99.2 [95.8 to 100.0] | 77.6 [65.8 to 86.9]
  Serotype 7F: number analyzed (Participants) | 72 | 176 | 71 | 127 | 76 | 131 | 67
  Serotype 7F | 100.0 [95.0 to 100.0] | 99.4 [96.9 to 100.0] | 4.2 [0.9 to 11.9] | 98.4 [94.4 to 99.8] | 21.1 [12.5 to 31.9] | 99.2 [95.8 to 100.0] | 37.3 [25.8 to 50.0]
  Serotype 9V: number analyzed (Participants) | 72 | 176 | 72 | 127 | 76 | 131 | 67
  Serotype 9V | 100.0 [95.0 to 100.0] | 98.3 [95.1 to 99.6] | 31.9 [21.4 to 44.0] | 99.2 [95.7 to 100.0] | 40.8 [29.6 to 52.7] | 100.0 [97.2 to 100.0] | 59.7 [47.0 to 71.5]
  Serotype 14 | 97.2 [90.3 to 99.7] | 99.4 [96.9 to 100.0] | 6.9 [2.3 to 15.5] | 98.4 [94.4 to 99.8] | 22.1 [13.4 to 33.0] | 100.0 [97.2 to 100.0] | 41.8 [29.8 to 54.5]
  Serotype 18C: number analyzed (Participants) | 72 | 176 | 72 | 127 | 77 | 131 | 66
  Serotype 18C | 100.0 [95.0 to 100.0] | 97.7 [94.3 to 99.4] | 5.6 [1.5 to 13.6] | 98.4 [94.4 to 99.8] | 15.6 [8.3 to 25.6] | 100.0 [97.2 to 100.0] | 40.9 [29.0 to 53.7]
  Serotype 19A | 100.0 [95.0 to 100.0] | 100.0 [97.9 to 100.0] | 63.9 [51.7 to 74.9] | 100.0 [97.1 to 100.0] | 90.9 [82.2 to 96.3] | 100.0 [97.2 to 100.0] | 94.0 [85.4 to 98.3]
  Serotype 19F | 98.6 [92.5 to 100.0] | 98.9 [96.0 to 99.9] | 29.2 [19.0 to 41.1] | 97.6 [93.3 to 99.5] | 44.2 [32.8 to 55.9] | 100.0 [97.2 to 100.0] | 70.1 [57.7 to 80.7]
  Serotype 23F: number analyzed (Participants) | 72 | 176 | 71 | 127 | 77 | 131 | 67
  Serotype 23F | 95.8 [88.3 to 99.1] | 95.5 [91.2 to 98.0] | 14.1 [7.0 to 24.4] | 97.6 [93.3 to 99.5] | 26.0 [16.6 to 37.2] | 96.9 [92.4 to 99.2] | 52.2 [39.7 to 64.6]

12. Secondary Outcome: Percentage of Participants Achieving Serotype-specific Pneumococcal OPA Titer ≥ Lower Limit of Quantitation (LLOQ) for 1 Month After the Last Vaccination in Cohorts 2,3,4 (13vPnC and Hib Vaccine) and 1 Month After the Infant Series in Cohort 1 (13vPnC).
Description: Serotype-specific OPA titers to the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in a randomly selected subset of about 50 participants receiving 13vPnC from the blood samples taken 1 month after the infant series in Cohort 1 and the last vaccination (13vPnC or Hib vaccine) in each of the 3 cohorts.
Time Frame: Cohort 1: 1 month after the 3rd dose of 13vPnC. Cohorts 2, 3, 4: 1 month after the last dose of 13vPnC and Hib Vaccine.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Cohort 1_Infant Series: Proportion of participants achieving serotype-specific pneumococcal OPA titer ≥ LLOQ for 1 month after infant series in Cohort 1.
- Cohort 2_13vPnC: Proportion of participants achieving serotype-specific pneumococcal OPA titer ≥ LLOQ for 1 month after the last dose of 13vPnC in Cohort 2.
- Cohort 2_Hib Vaccine: Proportion of participants achieving serotype-specific pneumococcal OPA titer ≥ LLOQ for 1 month after the last dose of Hib vaccine in Cohort 2.
- Cohort 3_13vPnC: Proportion of participants achieving serotype-specific pneumococcal OPA titer ≥ LLOQ for 1 month after the last dose of 13vPnC in Cohort 3.
- Cohort 3_Hib Vaccine: Proportion of participants achieving serotype-specific pneumococcal OPA titer ≥ LLOQ for 1 month after the last dose of Hib vaccine in Cohort 3.
- Cohort 4_13vPnC: Proportion of participants achieving serotype-specific pneumococcal OPA titer ≥ LLOQ for 1 month after the last dose of 13vPnC in Cohort 4.
- Cohort 4_Hib Vaccine: Proportion of participants achieving serotype-specific pneumococcal OPA titer ≥ LLOQ for 1 month after the last dose of Hib vaccine in Cohort 4.
Arm/Group | Cohort 1_Infant Series | Cohort 2_13vPnC | Cohort 2_Hib Vaccine | Cohort 3_13vPnC | Cohort 3_Hib Vaccine | Cohort 4_13vPnC | Cohort 4_Hib Vaccine
Number analyzed (Participants) | 37 | 87 | 34 | 78 | 42 | 71 | 36
Percentage of Participants
  Serotype 1 | 100.0 [90.5 to 100.0] | 96.6 [90.3 to 99.3] | 5.9 [0.7 to 19.7] | 96.2 [89.2 to 99.2] | 7.1 [1.5 to 19.5] | 95.8 [88.1 to 99.1] | 5.6 [0.7 to 18.7]
  Serotype 3 | 100.0 [90.5 to 100.0] | 100.0 [95.8 to 100.0] | 29.4 [15.1 to 47.5] | 100.0 [95.4 to 100.0] | 38.1 [23.6 to 54.4] | 100.0 [94.9 to 100.0] | 80.6 [64.0 to 91.8]
  Serotype 4 | 100.0 [90.5 to 100.0] | 100.0 [95.8 to 100.0] | 23.5 [10.7 to 41.2] | 100.0 [95.4 to 100.0] | 23.8 [12.1 to 39.5] | 100.0 [94.9 to 100.0] | 55.6 [38.1 to 72.1]
  Serotype 5 | 100.0 [90.5 to 100.0] | 100.0 [95.8 to 100.0] | 14.7 [5.0 to 31.1] | 100.0 [95.4 to 100.0] | 4.8 [0.6 to 16.2] | 98.6 [92.4 to 100.0] | 11.1 [3.1 to 26.1]
  Serotype 6A | 100.0 [90.5 to 100.0] | 100.0 [95.8 to 100.0] | 14.7 [5.0 to 31.1] | 100.0 [95.4 to 100.0] | 31.0 [17.6 to 47.1] | 100.0 [94.9 to 100.0] | 80.6 [64.0 to 91.8]
  Serotype 6B | 100.0 [90.5 to 100.0] | 94.3 [87.1 to 98.1] | 11.8 [3.3 to 27.5] | 98.7 [93.1 to 100.0] | 35.7 [21.6 to 52.0] | 100.0 [94.9 to 100.0] | 80.6 [64.0 to 91.8]
  Serotype 7F | 100.0 [90.5 to 100.0] | 100.0 [95.8 to 100.0] | 61.8 [43.6 to 77.8] | 100.0 [95.4 to 100.0] | 90.5 [77.4 to 97.3] | 100.0 [94.9 to 100.0] | 100.0 [90.3 to 100.0]
  Serotype 9V | 100.0 [90.5 to 100.0] | 100.0 [95.8 to 100.0] | 41.2 [24.6 to 59.3] | 100.0 [95.4 to 100.0] | 76.2 [60.5 to 87.9] | 100.0 [94.9 to 100.0] | 97.2 [85.5 to 99.9]
  Serotype 14 | 100.0 [90.5 to 100.0] | 100.0 [95.8 to 100.0] | 41.2 [24.6 to 59.3] | 100.0 [95.4 to 100.0] | 45.2 [29.8 to 61.3] | 100.0 [94.9 to 100.0] | 83.3 [67.2 to 93.6]
  Serotype 18C | 100.0 [90.5 to 100.0] | 98.9 [93.8 to 100] | 14.7 [5.0 to 31.1] | 98.7 [93.1 to 100.0] | 21.4 [10.3 to 36.8] | 100.0 [94.9 to 100.0] | 52.8 [35.5 to 69.6]
  Serotype 19A | 100.0 [90.5 to 100.0] | 100.0 [95.8 to 100.0] | 26.5 [12.9 to 44.4] | 100.0 [95.4 to 100.0] | 47.6 [32.0 to 63.6] | 100.0 [94.9 to 100.0] | 83.3 [67.2 to 93.6]
  Serotype 19F | 97.3 [85.8 to 99.9] | 100.0 [95.8 to 100.0] | 17.6 [6.8 to 34.5] | 100.0 [95.4 to 100.0] | 26.2 [13.9 to 42.0] | 100.0 [94.9 to 100.0] | 63.9 [46.2 to 79.2]
  Serotype 23F | 97.3 [85.8 to 99.9] | 95.4 [88.6 to 98.7] | 35.3 [19.7 to 53.5] | 96.2 [89.2 to 99.2] | 33.3 [19.6 to 49.5] | 97.2 [90.2 to 99.7] | 72.2 [54.8 to 85.8]

13. Secondary Outcome: Number of Participants With AE From the Signing of the ICD to 1 Month After the Infant Series in Cohort 1
Description: as for outcome 5
Time Frame: From the signing of ICD to 1 month after the 3rd dose of 13vPnC in Cohort 1.
Population: The safety population included all participants who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1_Infant Series
Number analyzed (Participants) | 125
Participants | 14

14. Secondary Outcome: Number of Participants With NDCMCs From 1 Month After Vaccination 3 to Vaccination 4 in Cohort 1
Description: Number of Participants With NDCMCs from 1 month after vaccination 3 to vaccination 4 in Cohort 1. An NDCMC was defined as a disease or medical condition that was not identified prior to study start and was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: From 1 month after Vaccination 3 to Vaccination 4.
Population: The safety population were participants who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1_Infant Series
Number analyzed (Participants) | 125
Participants | 0

15. Secondary Outcome: Number of Participants With AE From Toddler Dose Until 1 Month After the Toddler Dose in Cohort 1
Description: Number of Participants With AEs from vaccination 4 to 1 month after vaccination 4 in Cohort 1. An AE was any untoward medical occurrence in a study participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage.
Time Frame: From Vaccination 4 to 1 month after Vaccination 4 in Cohort 1.
Population: The safety population were participants who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1_ Toddler Dose: Participants vaccinated 4 doses of 13vPnC (single intramuscular injection): Vaccination 1 (Visit 1): 42 to 56 days of age; Vaccination 2 (Visit 2): 42 to 70 days after Visit 1; Vaccination 3 (Visit 3): 42 to 70 days after Visit 2; Vaccination 4: 365 to 455 days of age.
Arm/Group | Cohort 1_ Toddler Dose
Number analyzed (Participants) | 90
Participants | 5

16. Secondary Outcome: Number of Participants With NDCMCs From 1 Month to 6 Months After the Toddler Dose in Cohort 1
Description: Number of Participants With NDCMCs from 1 month after vaccination 4 to 6 months after vaccination 4 in Cohort 1. An NDCMC was defined as a disease or medical condition that was not identified prior to study start and was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: From 1 month to 6 months (5 months) after Vaccination 4 in Cohort 1.
Population: The safety population were participants who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 _Toddler Dose: Participants vaccinated 4 doses of 13vPnC (single intramuscular injection): Vaccination 1 (Visit 1): 42 to 56 days of age; Vaccination 2 (Visit 2): 42 to 70 days after Visit 1; Vaccination 3 (Visit 3): 42 to 70 days after Visit 2; Vaccination 4: 365 to 455 days of age.
Arm/Group | Cohort 1 _Toddler Dose
Number analyzed (Participants) | 90
Participants | 0

17. Secondary Outcome: Number of Participants With SAEs From the Signing of the ICD to 6 Months After the Toddler Dose in Cohort 1
Description: Number of Participants With SAEs from the signing of the ICD to 6 months after vaccination 4. An SAE was any untoward medical occurrence at any dose that resulted in death, was life-threatening (immediate risk of death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect or considered to be an important medical event.
Time Frame: From the Signing of the ICD to 6 Months After the Vaccination 4.
Population: The safety population were participants who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 125
Participants | 9

18. Secondary Outcome: Serotype-specific IgG GMCs for Each of the Pneumococcal Serotypes in Cohort 1 at 12, 24, 36 and 48 Months After Last Vaccination in Cohort 1 (Infant Series)
Description: Serotype-specific IgG concentrations to the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in all participants from the blood samples taken after last vaccination in Cohort 1. GMC and corresponding 2-sided 95% CI were evaluated. GMs were calculated using all participants with available data for the specified blood draw.
Time Frame: Cohort 1 (infant series): 12, 24, 36 and 48 Months After Last Vaccination in Cohort 1
Population: Evaluable analysis set was analyzed. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable at specific rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram/milliliter
Arm/Group | Cohort 1_Infant Series
Number analyzed (Participants) | 75
Microgram/milliliter
  Serotype 1: 12 Months After Last Vaccination in Cohort 1 | 1.35 [1.10 to 1.65]
  Serotype 1: 24 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 70
  Serotype 1: 24 Months After Last Vaccination in Cohort 1 | 0.88 [0.75 to 1.03]
  Serotype 1: 36 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 67
  Serotype 1: 36 Months After Last Vaccination in Cohort 1 | 0.77 [0.67 to 0.90]
  Serotype 1: 48 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 65
  Serotype 1: 48 Months After Last Vaccination in Cohort 1 | 0.79 [0.69 to 0.91]
  Serotype 3: 12 Months After Last Vaccination in Cohort 1 | 0.27 [0.24 to 0.31]
  Serotype 3: 24 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 70
  Serotype 3: 24 Months After Last Vaccination in Cohort 1 | 0.22 [0.17 to 0.28]
  Serotype 3: 36 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 67
  Serotype 3: 36 Months After Last Vaccination in Cohort 1 | 0.18 [0.14 to 0.21]
  Serotype 3: 48 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 65
  Serotype 3: 48 Months After Last Vaccination in Cohort 1 | 0.19 [0.13 to 0.26]
  Serotype 4: 12 Months After Last Vaccination in Cohort 1 | 1.10 [0.90 to 1.35]
  Serotype 4: 24 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 70
  Serotype 4: 24 Months After Last Vaccination in Cohort 1 | 0.54 [0.41 to 0.71]
  Serotype 4: 36 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 67
  Serotype 4: 36 Months After Last Vaccination in Cohort 1 | 0.58 [0.45 to 0.75]
  Serotype 4: 48 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 65
  Serotype 4: 48 Months After Last Vaccination in Cohort 1 | 0.32 [0.23 to 0.44]
  Serotype 5: 12 Months After Last Vaccination in Cohort 1 | 1.56 [1.35 to 1.81]
  Serotype 5: 24 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 70
  Serotype 5: 24 Months After Last Vaccination in Cohort 1 | 1.03 [0.91 to 1.17]
  Serotype 5: 36 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 67
  Serotype 5: 36 Months After Last Vaccination in Cohort 1 | 1.03 [0.91 to 1.17]
  Serotype 5: 48 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 65
  Serotype 5: 48 Months After Last Vaccination in Cohort 1 | 1.19 [1.05 to 1.34]
  Serotype 6A: 12 Months After Last Vaccination in Cohort 1 | 2.10 [1.71 to 2.59]
  Serotype 6A: 24 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 70
  Serotype 6A: 24 Months After Last Vaccination in Cohort 1 | 1.40 [1.12 to 1.74]
  Serotype 6A: 36 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 67
  Serotype 6A: 36 Months After Last Vaccination in Cohort 1 | 2.79 [2.04 to 3.80]
  Serotype 6A: 48 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 65
  Serotype 6A: 48 Months After Last Vaccination in Cohort 1 | 3.06 [2.30 to 4.06]
  Serotype 6B: 12 Months After Last Vaccination in Cohort 1 | 2.40 [1.94 to 2.95]
  Serotype 6B: 24 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 70
  Serotype 6B: 24 Months After Last Vaccination in Cohort 1 | 2.12 [1.69 to 2.66]
  Serotype 6B: 36 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 67
  Serotype 6B: 36 Months After Last Vaccination in Cohort 1 | 3.29 [2.57 to 4.21]
  Serotype 6B: 48 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 65
  Serotype 6B: 48 Months After Last Vaccination in Cohort 1 | 3.73 [2.95 to 4.71]
  Serotype 7F: 12 Months After Last Vaccination in Cohort 1 | 1.55 [1.31 to 1.82]
  Serotype 7F: 24 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 70
  Serotype 7F: 24 Months After Last Vaccination in Cohort 1 | 0.77 [0.67 to 0.88]
  Serotype 7F: 36 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 67
  Serotype 7F: 36 Months After Last Vaccination in Cohort 1 | 0.62 [0.56 to 0.70]
  Serotype 7F: 48 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 65
  Serotype 7F: 48 Months After Last Vaccination in Cohort 1 | 0.53 [0.41 to 0.68]
  Serotype 9V: 12 Months After Last Vaccination in Cohort 1 | 1.32 [1.11 to 1.57]
  Serotype 9V: 24 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 70
  Serotype 9V: 24 Months After Last Vaccination in Cohort 1 | 0.88 [0.74 to 1.04]
  Serotype 9V: 36 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 67
  Serotype 9V: 36 Months After Last Vaccination in Cohort 1 | 0.84 [0.72 to 0.99]
  Serotype 9V: 48 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 65
  Serotype 9V: 48 Months After Last Vaccination in Cohort 1 | 0.95 [0.78 to 1.16]
  Serotype 14: 12 Months After Last Vaccination in Cohort 1 | 2.77 [2.30 to 3.34]
  Serotype 14: 24 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 70
  Serotype 14: 24 Months After Last Vaccination in Cohort 1 | 2.03 [1.52 to 2.70]
  Serotype 14: 36 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 67
  Serotype 14: 36 Months After Last Vaccination in Cohort 1 | 2.49 [1.76 to 3.51]
  Serotype 14: 48 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 64
  Serotype 14: 48 Months After Last Vaccination in Cohort 1 | 2.14 [1.34 to 3.42]
  Serotype 18C: 12 Months After Last Vaccination in Cohort 1 | 1.24 [1.07 to 1.43]
  Serotype 18C: 24 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 70
  Serotype 18C: 24 Months After Last Vaccination in Cohort 1 | 0.72 [0.58 to 0.89]
  Serotype 18C: 36 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 67
  Serotype 18C: 36 Months After Last Vaccination in Cohort 1 | 0.67 [0.54 to 0.81]
  Serotype 18C: 48 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 65
  Serotype 18C: 48 Months After Last Vaccination in Cohort 1 | 0.60 [0.47 to 0.78]
  Serotype 19A: 12 Months After Last Vaccination in Cohort 1 | 2.92 [2.29 to 3.74]
  Serotype 19A: 24 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 70
  Serotype 19A: 24 Months After Last Vaccination in Cohort 1 | 3.52 [2.68 to 4.63]
  Serotype 19A: 36 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 67
  Serotype 19A: 36 Months After Last Vaccination in Cohort 1 | 6.39 [4.79 to 8.51]
  Serotype 19A: 48 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 65
  Serotype 19A: 48 Months After Last Vaccination in Cohort 1 | 7.53 [6.14 to 9.22]
  Serotype 19F: 12 Months After Last Vaccination in Cohort 1 | 2.88 [2.32 to 3.57]
  Serotype 19F: 24 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 70
  Serotype 19F: 24 Months After Last Vaccination in Cohort 1 | 2.73 [2.01 to 3.72]
  Serotype 19F: 36 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 67
  Serotype 19F: 36 Months After Last Vaccination in Cohort 1 | 4.06 [2.92 to 5.66]
  Serotype 19F: 48 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 65
  Serotype 19F: 48 Months After Last Vaccination in Cohort 1 | 3.51 [2.56 to 4.80]
  Serotype 23F: 12 Months After Last Vaccination in Cohort 1 | 2.14 [1.76 to 2.59]
  Serotype 23F: 24 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 70
  Serotype 23F: 24 Months After Last Vaccination in Cohort 1 | 1.72 [1.44 to 2.04]
  Serotype 23F: 36 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 67
  Serotype 23F: 36 Months After Last Vaccination in Cohort 1 | 1.92 [1.58 to 2.34]
  Serotype 23F: 48 Months After Last Vaccination in Cohort 1: number analyzed (Participants) | 65
  Serotype 23F: 48 Months After Last Vaccination in Cohort 1 | 2.15 [1.75 to 2.63]

ADVERSE EVENTS:
Time Frame: AE for Cohort 1: from the signing of the ICD to 1 month after Vaccination 3 and from Vaccination 4 to 1 month after Vaccination 4. AE for Cohorts 2,3,4: from the signing of the ICD to 1 month after the last study vaccination. SAE for Cohort 1,2,3,4: From the signing of the ICD to 6 months after the last study vaccination. See below for detailed vaccination timepoints in each cohort.
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. The safety population were participants who received at least 1 dose of the investigational product.
Groups:
- Cohort 1: Participants vaccinated 4 doses of 13vPnC (single intramuscular injection): Vaccination 1 (Visit 1): 42 to 56 days of age; Vaccination 2 (Visit 2): 42 to 70 days after Visit 1; Vaccination 3: 42 to 70 days after Visit 2; Vaccination 4: 365 to 455 days of age.
- Cohort 2_Hib Vaccine: Participants vaccinated 2 doses of Hib Vaccine (single intramuscular injection): Vaccination 1 (Visit 1): 7 to <12 months of age; Vaccination 2: at least 28 days after Visit 1;
- Cohort 3_Hib Vaccine: Participants vaccinated 1 dose of Hib vaccine (single intramuscular injection): Vaccination 1: >=1 to <2 years of age;
Arm/Group | Cohort 1 | Cohort 2_13vPnC | Cohort 2_Hib Vaccine | Cohort 3_13vPnC | Cohort 3_Hib Vaccine | Cohort 4_13vPnC | Cohort 4_Hib Vaccine
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/236 | 0/117 | 0/165 | 0/83 | 0/138 | 0/68
Serious Adverse Events (participants affected / at risk) | 9/125 | 5/236 | 1/117 | 2/165 | 0/83 | 2/138 | 1/68
Other Adverse Events (participants affected / at risk) | 13/125 | 182/236 | 74/117 | 99/165 | 26/83 | 66/138 | 29/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=125) | Cohort 2_13vPnC (N=236) | Cohort 2_Hib Vaccine (N=117) | Cohort 3_13vPnC (N=165) | Cohort 3_Hib Vaccine (N=83) | Cohort 4_13vPnC (N=138) | Cohort 4_Hib Vaccine (N=68)
Pneumonia (Infections and infestations) | 7 | 1 | 0 | 1 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=125) | Cohort 2_13vPnC (N=236) | Cohort 2_Hib Vaccine (N=117) | Cohort 3_13vPnC (N=165) | Cohort 3_Hib Vaccine (N=83) | Cohort 4_13vPnC (N=138) | Cohort 4_Hib Vaccine (N=68)
Pyrexia (General disorders) | 3 | 31 | 13 | 8 | 1 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 22 | 6 | 5 | 0 | 3 | 0
Pyrexia (FEVER) (General disorders) | 0 | 121 | 37 | 55 | 16 | 20 | 16
Swelling (SWELLING) (General disorders) | 0 | 38 | 5 | 21 | 3 | 27 | 16
Tenderness (TENDERNESS) (General disorders) | 0 | 18 | 2 | 18 | 3 | 26 | 15
Decreased appetite (DECREASED APPETITE) (Metabolism and nutrition disorders) | 0 | 6 | 2 | 13 | 3 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 22 | 9 | 1 | 0 | 0 | 0
Erythema (REDNESS) (Skin and subcutaneous tissue disorders) | 1 | 68 | 27 | 42 | 10 | 36 | 15
Fatigue (FATIGUE) (General disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 6
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 1 | 0 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (VOMITING) (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 2 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 3 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Viral rash (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Hand-foot-and -mouth disease (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersomnia (INCREASED SLEEP) (Nervous system disorders) | 0 | 5 | 0 | 3 | 3 | 0 | 0
Headache (HEADACHE) (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Irritability (IRRITABILITY) (Psychiatric disorders) | 0 | 3 | 1 | 7 | 2 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 1
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT03574389/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT03574389/SAP_001.pdf